CLINICAL TRIAL: NCT06137469
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Crossover Study to Assess the Effect of Multiple Subcutaneous Injections of SHR20004 in Healthy Subjects on Gastric Emptying
Brief Title: Assessment of Gastric Emptying by SHR20004 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SHR20004-106
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: This study is a single-center, randomized, double-blind, placebo-controlled, crossover study. Healthy subjects were randomly assigned to receive SHR20004 or placebo treatment. In the group receiving SHR20004, the pharmacokinetic changes of acetaminophen were compared before and after treatment with SHR20004.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetaminophen+SHR20004 (Experimental)
  Interventions: Drug: Acetaminophen/SHR20004
- Acetaminophen+Placebo (Experimental)
  Interventions: Drug: Acetaminophen/Placebo

INTERVENTIONS:
Drug: Acetaminophen/SHR20004 — SHR20004 was administered by titration, with all subjects starting on Day 4 with an initial dose of 0.03 mg/d of SHR20004 or placebo, with the dose being increased by 0.03 mg/d per week. The dose was increased to 0.15 mg/d and then maintained for 5 days.
  Arms: Acetaminophen+SHR20004
Drug: Acetaminophen/Placebo — Placebo was administered by titration, with all subjects starting on Day 4 with an initial dose of 0.03 mg/d of SHR20004 or placebo, with the dose being increased by 0.03 mg/d per week. The dose was increased to 0.15 mg/d and then maintained for 5 days.
  Arms: Acetaminophen+Placebo

SUMMARY:
The purpose of this study is to investigate the impact of SHR20004 on the pharmacokinetic (PK) characteristics of acetaminophen in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form before participating in activities related to this trial and be able to understand the procedures and methods of the trial. Be willing to strictly follow the clinical trial protocol to complete the trial.
2. Healthy males or females aged 18-55 years (inclusive, as of signing the informed consent form).
3. Body mass index (BMI) between 19 and 28 kg/m2 (inclusive), with a weight ≥ 50 kg.
4. Have not used GLP-1 or its analogs, DPP Ⅳ inhibitors or its analogs, or other glucose-lowering drugs.

Exclusion Criteria:

-

1. Subjects with any of the following conditions or medical history:

1. Any clinical disease that the investigator determines may affect the safety or results of the study.
2. Diagnosed with diabetes according to the WHO guidelines for the diagnosis and management of diabetes.
3. A history of thyroid cancer or family history of thyroid cancer, a history of pancreatitis, or symptomatic gallstones.
4. History of severe systemic infection within 1 month of screening.
5. History of severe cardiovascular disease, including decompensated heart failure (NYHA class III or IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, persistent and clinically significant arrhythmia, or history of coronary artery bypass surgery or percutaneous coronary intervention.
6. Subjects with clinically significant abnormal thyroid function at screening.
7. Prolonged QTcF interval on screening or baseline ECG (male > 450 ms, female > 470 ms), or other clinically significant abnormalities that may result in a significant safety risk for the subjects.
8. Subjects with severe mental disorders.

2. Use of prescription drugs (topical eye/ nasal drops and ointments are allowed) and over-the-counter drugs, food supplements, vitamins, and Chinese herbs within 2 weeks before the start of treatment (routine vitamins are allowed).

3. Any of the following:

1. A history of recurrent or severe drug-food allergies, or known or suspected allergy to any component of the investigational drug.
2. Participation in any drug clinical trial within the past 3 months (defined as receiving trial drug treatment).
3. Consumption of more than 14 standard units of alcohol per week (1 standard unit contains 14 g of alcohol, such as 360 mL of beer or 45 mL of alcohol with a 40% alcohol content or 150 mL of wine) within the past 1 year, or a positive breath alcohol test.
4. A history of smoking (≥5 cigarettes per day for the past 1 year) or a history of smoking in the past 1 year; subjects who cannot or are unwilling to abstain from smoking during the study period, or subjects who cannot use nicotine gum or transdermal nicotine patches.
5. Long-term or consumption within the past 48 hours of coffee, tea, chocolate, or soft drinks that contain methylxanthines (theophylline, caffeine, or theobromine), such as Coca-Cola.
6. Participation in intense exercise within the past 48 hours, such as weightlifting, sprinting, long-distance running, cycling, swimming, or soccer.
7. Known or suspected history of drug abuse or a positive urine drug screening test during screening.
8. Blood donation of ≥400 mL within the past 3 months or subjects with a bleeding event of ≥400 mL within the past 3 months, such as major surgery or trauma.
9. Positive serology for hepatitis B surface antigen (HBsAg), hepatitis C (HCV), syphilis, or human immunodeficiency virus (HIV) antibodies.
10. Subjects who are assessed by the investigator as having poor compliance or arm vein condition that cannot allow blood to be drawn, or subjects with a history of fainting or dizziness with needles.
11. Pregnant and lactating women, or male and female subjects who are of childbearing age and do not wish to use effective contraception for 2 weeks after the last dose of study medication.
12. Subjects who, in the opinion of the investigator, have any other condition that could interfere with the evaluation of the trial results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of acetaminophen after a single dose of 1.0 g was measured after administration of the standardized meal.：(AUC0-300min) | Based on pre-dose to 300 min post-dose sampling times on Day 1 and Day 31

SECONDARY OUTCOMES:
Pharmacokinetics parameters of acetaminophen after a single dose of 1.0 g was measured after administration of the standardized meal.： (AUC0-60min) | Based on pre-dose to 300 min post-dose sampling times on Day 1 and Day 31
Pharmacokinetics parameters of acetaminophen after a single dose of 1.0 g was measured after administration of the standardized meal.： (AUC0-60min/AUC0-300min) | Based on pre-dose to 300 min post-dose sampling times on Day 1 and Day 31
Pharmacokinetics parameters of acetaminophen after a single dose of 1.0 g was measured after administration of the standardized meal.： (Cmax) | Based on pre-dose to 300 min post-dose sampling times on Day 1 and Day 31
Pharmacokinetics parameters of acetaminophen after a single dose of 1.0 g was measured after administration of the standardized meal.： (Tmax) | Based on pre-dose to 300 min post-dose sampling times on Day 1 and Day 31
Pharmacokinetics parameters of acetaminophen after a single dose of 1.0 g was measured after administration of the standardized meal.： (t1/2) | Based on pre-dose to min post-dose sampling times on Day 1 and Day 31
Pharmacokinetics parameters of acetaminophen after a single dose of 1.0 g was measured after administration of the standardized meal.： (CL/F) | Based on pre-dose to 300 min post-dose sampling times on Day 1 and Day 31
Pharmacokinetics parameters of acetaminophen after a single dose of 1.0 g was measured after administration of the standardized meal.： (Vz/F) | Based on pre-dose to 300 min post-dose sampling times on Day 1 and Day 31
Incidence and severity of AE/SAE/AESI. | Screening period up to Day 50
Electrocardiographic parameters Fridericia-corrected QT interval (QTcF) | Day 1 and Day 10 and Day 30 and Day 36
  Mean QTcF as measured based on triplicate electrocardiograms extracted from continuous 12-lead Holter monitor recordings.
Delta QTcF | Day 1 and Day 10 and Day 30 and Day 36
  Mean change from baseline in QTcF as measured based on triplicate electrocardiograms extracted from continuous 12-lead Holter monitor recordings after study drug intake.
Double-delta QTcF (ΔΔQTcF) | Day 1 and Day 10 and Day 30 and Day 36
  Mean change from baseline and placebo in QTcF as measured based on triplicate electrocardiograms extracted from continuous 12-lead Holter monitor recordings after study drug intake.
Concentration-delta QTcF Correlation | Day 1 and Day 10 and Day 30 and Day 36
  Correlation between SHR20004 plasma concentration and delta QTcF based on appropriate regression model.
Concentration-double-delta QTcF Correlation | Day 1 and Day 10 and Day 30 and Day 36
  Correlation between SHR20004 plasma concentration and double-delta QTcF based on appropriate regression model.
Immunogenicity indicators: anti-Noiiglutide antibodies | Start of treatment up to Day 50

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided